CLINICAL TRIAL: NCT06256484
Title: A Phase 1 Study to Evaluate the Safety and Preliminary Efficacy of ATA3219, Allogeneic Anti-CD19 Chimeric Antigen Receptor T-cell Therapy, in Subjects With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: A Study to Evaluate the Safety and Preliminary Efficacy of ATA3219 in Participants With Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Financial reasons
Sponsor: Atara Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATA3219-NHL-103
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Relapsed/Refractory B-cell Non-Hodgkin Lymphoma
Keywords: B-cell non-Hodgkin Lymphoma; Anaplastic lymphoma kinase; Epstein-Barr virus (EBV); Mantle cell lymphoma (MCL); Follicular lymphoma (FL); Diffuse Large B-cell Lymphoma (DLBCL); Large B-cell lymphoma (LBCL)
MeSH Terms: conditions — Lymphoma, B-Cell; Epstein-Barr Virus Infections; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ATA3219 Dose Level 1 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 1 on Day 1.
  Interventions: Drug: ATA3219
- ATA3219 Dose Level 2 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 2 on Day 1.
  Interventions: Drug: ATA3219
- ATA3219 Dose Level 3 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 3 on Day 1.
  Interventions: Drug: ATA3219
- ATA3219 Dose Level 4 (Experimental): Participants will receive a single IV infusion of ATA3219 Dose Level 4 on Day 1.
  Interventions: Drug: ATA3219

INTERVENTIONS:
Drug: ATA3219 — ATA3219 is allogeneic anti-CD19 chimeric antigen receptor T-cell, administered intravenously on Day 1.

SUMMARY:
The purpose of this study is to evaluate the safety and preliminary efficacy of ATA3219 in participants with relapsed/refractory (R/R) B-cell non-Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
This is a phase 1, open-labeled study to evaluate the safety and preliminary efficacy of ATA3219 (as monotherapy) in participants with NHL. During dose escalation, participants with R/R large B-cell lymphoma (LBCL), follicular lymphoma (FL), or mantle cell lymphoma (MCL) may be enrolled sequentially. Up to 4 dose levels will be explored in dose escalation. Prior to undergoing any screening procedure, prospective participants must undergo the ATA3219 inventory check assessments to ensure availability of an appropriate partially human leukocyte antigen-matched ATA3219 lot. Before administration of ATA3219, participants will receive conditioning chemotherapy within 7 days of enrollment. Participants will be hospitalized for at least 1 week to receive ATA3219, which will be administered by intravenous (IV) infusion on Day 1 in a staggered manner to allow appropriate safety monitoring. Four different dose levels will be studied in a sequential manner, and a lower dose level may be added, if needed. At least 3 and up to 6 dose-limiting toxicity (DLT)-evaluable participants, those who complete the 28-day DLT observation period, will be assessed at each dose level. Disease response will be assessed on Day 28 (+ 5 days) following each dose of ATA3219 by the investigator using the Lugano criteria (Cheson 2014). Participants who achieve complete response (CR) or progressive disease at Day 28 will enter the 24-month follow-up period. Participants who achieve partial response (PR), stable disease, or those who relapse within 12 months of the ATA3219 dose, may be considered for the second dose of ATA3219 per protocol. A third and final dose of ATA3219 may also be considered as per protocol.

After recommended phase 2 dose (RP2D) has been determined in the dose escalation stage, additional participants may be enrolled in 2 expansion cohorts (CD19-directed naive and prior CD19-directed therapy), opened at sponsor discretion and dosed at the proposed RP2D.

After treatment is completed or discontinued, participants will be followed for response and safety for up to 24 months from the last dose of ATA3219. After 2 years, a separate long-term follow-up study will be conducted to follow participants for up to a total of 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, R/R, B-cell NHL according to the 2022 revision of the World Health Organization classification of lymphoid neoplasms [Alaggio 2022] defined as any of the following:

  1. LBCL
  2. FL Grade 3b
  3. MCL
* The following criteria apply for details of prior treatment/therapy: R/R to at least 2 lines of therapy; if the most recent line of therapy was autologous hematologic cell transplant (HCT), relapse within 12 months of the transplant.
* Measurable disease by scan (diagnostic positron emission tomography-positive and/or computed tomography-measurable) as per Lugano Classification [Cheson 2014]. Magnetic resonance imaging may be used when computed tomography with contrast is contraindicated or when mandated by local practice.
* If sufficient archival material is not available from the latest relapse, a new tumor biopsy is required any time during screening, prior to conditioning chemotherapy.
* Participants who have received prior CD19-directed therapy as the prior line of therapy:

  1. must have achieved either a CR or partial response as a best response and maintained the response for ≥ 3 months after receiving CD19-directed treatment, and
  2. must still have CD19+ disease as determined by a local laboratory.
* Eastern Cooperative Oncology Group performance status ≤ 2
* Adequate organ function
* Written informed consent as per protocol.
* Participants are able to commit to the inpatient portion of the study, encompassing conditioning (if per the institution's standard practice), and frequent monitoring during Days 1-15, as well as remain within 1 hour travel time of the clinical site for 28 days after each infusion.

Exclusion Criteria:

* History of a human immunodeficiency virus infection or acute or chronic active hepatitis B or C infection.
* History or presence of clinically relevant central nervous system (CNS) pathology.
* Unresolved Grade 1-2 Immune effector cell-associated neurotoxicity syndrome (ICANS) or experienced Grade 3-4 ICANS from prior chimeric antigen receptor T-cell.
* Unresolved graft-versus-host disease (GvHD) or Grade 3-4 acute GvHD from any prior therapy or moderate to severe chronic GvHD from any prior therapy.
* History of any one of the following cardiovascular conditions: class III or IV heart failure as defined by the New York Heart Association [The Criteria Committee of the New York Heart Association 1994], cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically meaningful cardiac disease, within the past 6 months of study informed consent.
* History of malignancies, other than R/R NHL, unless the participant has been disease-free for ≥ 1 year (certain noninvasive malignancies are allowed).
* Active primary, CNS-only, or systemic plus CNS involvement by lymphoma, unless the CNS involvement has been effectively treated.
* Active autoimmune disorders or inflammatory conditions that require systemic immunosuppressive therapies, including therapeutic doses of steroids.
* Has received prior allogeneic HCT or prior solid organ transplant.
* Systemic bacterial, viral, fungal, or other infection that is untreated or unresponsive to appropriate treatment (or requires IV antibiotics at enrollment); participants must be afebrile for ≥ 48 hours. Prophylactic antibiotics, antivirals, and antifungals are permitted.
* Concurrent serious uncontrolled or unresolved medical condition, including any laboratory abnormality or psychiatric illness.
* The following therapies within defined periods prior to the conditioning regimen: therapeutic doses of corticosteroids (> 0.5 mg/kg/day of prednisone or equivalent), lymphodepleting chemotherapeutic agents, live attenuated vaccines, prior systemic cancer therapy, investigational agents, including approved drugs being used off label, autologous HCT, donor lymphocyte infusions, radiation, alemtuzumab.
* Female who is breastfeeding or pregnant.
* Inability or unwillingness to comply with study procedures.
* Unwilling to use protocol specified contraceptive methods.
* Life expectancy of ≤ 8 weeks.
* For participants being considered for retreatment: had a DLT with prior ATA3219 dose.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-09-06 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Treatment-emergent Adverse Events (TEAEs) | Day 1 through 90 days after the last dose of study drug
Incidence and Severity of Adverse Events of Special Interest (AESIs) | Day 1 through 90 days after the last dose of study drug
Number of Participants With Clinically Significant Changes in Laboratory Parameters | Day 1 through 90 days after the last dose of study drug
Incidence of Dose-limiting Toxicities (DLTs) | Day 1 through Day 28 of first dose
Maximum Tolerated dose (MTD) | Day 1 through Day 28 of first dose
Recommended Phase 2 Dose (RP2D) | Day 1 through Day 28 of first dose

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ATA3219 | Pre-dose Day 1 through 24 months after last dose on a defined schedule
Time to Reach Cmax of ATA3219 | Pre-dose Day 1 through 24 months after last dose on a defined schedule
Partial Area Under the Curve (pAUC) of ATA3219 | Pre-dose Day 1 through 24 months after last dose on a defined schedule
Last Observed Plasma Concentration (Clast) of ATA3219 | Pre-dose Day 1 through 24 months after last dose on a defined schedule
Time of Clast of ATA3219 | Pre-dose Day 1 through 24 months after last dose on a defined schedule
Terminal Half-life (T1/2) of ATA3219 | Pre-dose Day 1 through 24 months after last dose on a defined schedule
Objective Response Rate (ORR) | Screening (≤ 28 days before enrollment) through 24 months after last dose
Complete Response Rate (CRR) | Screening (≤ 28 days before enrollment) through 24 months after last dose
Time-to-response (TTR) | Screening (≤ 28 days before enrollment) through 24 months after last dose
Duration of Response (DOR) | Screening (≤ 28 days before enrollment) through 24 months after last dose
Progression-free Survival (PFS) | Screening (≤ 28 days before enrollment) through 24 months after last dose
Overall Survival (OS) | Screening (≤ 28 days before enrollment) through 24 months after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Aditi Mehta, DO, Study Director — Atara Biotherapeutics
Locations (6):
- United States (4):
  - AdventHealth Cancer Institute, Orlando, Florida
  - Norton Cancer Institute - Saint Matthews, Louisville, Kentucky
  - Sidney Kimmel Cancer Center - Jefferson Health, Philadelphia, Pennsylvania
  - University of Virgina, Charlottesville, Virginia
- Australia (2):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Fiona Stanley Hospital, Murdoch, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Alaggio R, Amador C, Anagnostopoulos I, Attygalle AD, Araujo IBO, Berti E, Bhagat G, Borges AM, Boyer D, Calaminici M, Chadburn A, Chan JKC, Cheuk W, Chng WJ, Choi JK, Chuang SS, Coupland SE, Czader M, Dave SS, de Jong D, Du MQ, Elenitoba-Johnson KS, Ferry J, Geyer J, Gratzinger D, Guitart J, Gujral S, Harris M, Harrison CJ, Hartmann S, Hochhaus A, Jansen PM, Karube K, Kempf W, Khoury J, Kimura H, Klapper W, Kovach AE, Kumar S, Lazar AJ, Lazzi S, Leoncini L, Leung N, Leventaki V, Li XQ, Lim MS, Liu WP, Louissaint A Jr, Marcogliese A, Medeiros LJ, Michal M, Miranda RN, Mitteldorf C, Montes-Moreno S, Morice W, Nardi V, Naresh KN, Natkunam Y, Ng SB, Oschlies I, Ott G, Parrens M, Pulitzer M, Rajkumar SV, Rawstron AC, Rech K, Rosenwald A, Said J, Sarkozy C, Sayed S, Saygin C, Schuh A, Sewell W, Siebert R, Sohani AR, Tooze R, Traverse-Glehen A, Vega F, Vergier B, Wechalekar AD, Wood B, Xerri L, Xiao W. The 5th edition of the World Health Organization Classification of Haematolymphoid Tumours: Lymphoid Neoplasms. Leukemia. 2022 Jul;36(7):1720-1748. doi: 10.1038/s41375-022-01620-2. Epub 2022 Jun 22. PMID 35732829